CLINICAL TRIAL: NCT05317728
Title: Randomized Controlled Study of Fluid Accommodating IOL Outcomes Versus Monofocal Control
Brief Title: Clinical Study of a Fluid Accommodating Intraocular Lens (IOL) Design
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: ILR286-E002
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cataract
Keywords: IOL; Intraocular lens
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Cohort 1 utilizes a parallel-group study design. Cohort 2 utilizes a single-group study design.
Who Masked: Participant, Outcomes Assessor
Masking Description: Cohort 1 is a subject and assessor-masked comparison. Cohort 2 does not utilize masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Cohort 1: BAL-FAIOL (Experimental): BAL-FAIOL IOL implanted in both eyes during cataract surgery (bilateral implantation)
  Interventions: Device: BAL-FAIOL IOL; Procedure: Cataract surgery
- Cohort 1: Monofocal (Active Comparator): Monofocal IOL implanted in both eyes during cataract surgery (bilateral implantation)
  Interventions: Device: Monofocal IOL; Procedure: Cataract surgery
- Cohort 2: BAL-FAIOL (Experimental): BAL-FAIOL IOL implanted in both eyes during cataract surgery (bilateral implantation)
  Interventions: Device: BAL-FAIOL IOL; Procedure: Cataract surgery

INTERVENTIONS:
Device: BAL-FAIOL IOL — Investigational implantable medical device intended for long-term use over the lifetime of the cataract subject
  Arms: Cohort 1: BAL-FAIOL; Cohort 2: BAL-FAIOL
Device: Monofocal IOL — Commercially available implantable medical device intended for long-term use over the lifetime of the cataract subject
  Other Names: AcrySof IQ monofocal IOL (SN60WF)
  Arms: Cohort 1: Monofocal
Procedure: Cataract surgery — Phacoemulsification with a clear cornea incision

SUMMARY:
The purpose of this clinical study is to evaluate the surgical, refractive, and visual outcomes with implantation of an investigational intraocular lens (IOL).

DETAILED DESCRIPTION:
In this study, eligible subjects will receive cataract surgery with IOL implantation in both eyes. IOL implantation in the second eye is intended to occur between 7 and 15 days after IOL implantation in the first eye. Subjects will be followed for 1 year after implantation.

This study will enroll 2 cohorts. Cohort 1 subjects will be randomized to receive either the test IOL (BAL-FAIOL) or the control IOL (Monofocal). Cohort 2 subjects will receive the test IOL only (BAL-FAIOL). Cohort 2 will follow Cohort 1.

This study will be conducted in Central America.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an Institutional Review Board / International Ethics Committee approved informed Consent form;
* Willing and able to attend all scheduled study visits as required by the protocol;
* Diagnosed with bilateral cataracts requiring removal by phacoemulsification with a clear corneal incision;
* Other protocol-specified inclusion criteria may apply.

Key Exclusion Criteria:

* Subjects taking medications that may affect accommodation;
* Clinically significant eye abnormalities as specified in the protocol;
* Previous eye surgery as specified in the protocol;
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Mean Photopic Monocular Best Corrected Distance Visual Acuity (BCDVA) (4 meters) | Month 6 post second eye implantation
  Distance visual acuity will be measured with correction in place for each eye individually using letter charts and recorded in logarithm Minimum Angle of Resolution (logMAR). This outcome measure is pre-specified for Cohort 1 and Cohort 2.
Cumulative Adverse Events, including Secondary Surgical Interventions (SSIs) | Up to Year 1
  The number of adverse events, including SSI's, will be calculated from time of implantation. This outcome measure is pre-specified for Cohort 1 BAL-FAIOL IOL only.
Cumulative Adverse Events, including Secondary Surgical Interventions (SSIs) - Cohort 2 | Up to Year 1
  The number of adverse events, including SSI's, will be calculated from time of implantation. The outcome measure is pre-specified for Cohort 2 only

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Surgical, Study Director — Alcon Research, LLC
Locations (6):
- Clinica 20/20, San José, Costa Rica
- Laser Center SA, Santo Domingo, Dominican Republic
- Mexico (3):
  - Centro de Retina Medica y Quirurgica SC, Zapopan, Jalisco
  - Asociación Para Evitar la Ceguera en México, Mexico City
  - Salauno Salud SAPI de CV, Mexico City
- Panama Eye Center, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No